CLINICAL TRIAL: NCT00612144
Title: A Multicenter, Randomized, Parallel-group, Open Study to Compare the Efficacy and Safety of Early Combination Therapy With Amaryl M to Metformin Uptitration in Type 2 DM Patients Inadequately Controlled on Metformin HCL
Brief Title: Study Comparing Efficacy and Safety of Amaryl M and Metformin Uptitraion to Type 2 DM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Responsible Party: Moon-Hwa Park, Head of Medical Affairs, Medical Affairs
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLIME_L_02861
Record Dates: First submitted 2008-01-07; First posted 2008-02-11 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — glimepiride; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Amaryl M group
  Interventions: Drug: Glimepiride/metformin fixed combination
- 2 (Active Comparator): Metformin group
  Interventions: Drug: Metformin HCl

INTERVENTIONS:
Drug: Glimepiride/metformin fixed combination — Amaryl M 1/250mg~4/1000mg bid for 12~26 weeks
  * Maintenance dose for 10 weeks after 2~14 weeks of dose titration
  * Dose titration according to titration algorithm based on daily mean SMBG
  Other Names: Amaryl M
  Arms: 1
Drug: Metformin HCl — Metformin HCl 500mg~1250mg bid for 12~26 weeks
  * Maintenance dose for 10 weeks after 2~14 weeks of dose titration
  * Dose titration according to titration algorithm based on daily mean SMBG
  Other Names: Diabex
  Arms: 2

SUMMARY:
The aim of this study is to compare the efficacy and safety of early combination therapy with Amaryl M with that of uptitration of metformin monotherapy in patients with type 2 DM inadequately controlled by prior monotherapy with metformin.

DETAILED DESCRIPTION:
Treatment algorithms for type 2 DM generally employ monotherapy as a first-line pharmacologic treatment option. Disease progression renders monotherapy less effective in controlling blood glucose over time, with approximately half of the patients requiring additional therapy by 3 years after diagnosis. As a result, the use of multiple pharmacologic agents to control blood glucose is well accepted.

In combination therapy, selection of suitable drug may be individualized depending on their health conditions. However, it is advisable to select drugs having different mechanism considering their complimentary action with each other. Therefore, sulfonylureas and metformin HCL is the best combination in which "insulin deficiency" and "insulin resistance", the basic two pathophysiologies in type 2 diabetes could be targeted. The efficacy and safety of the combination with sulfonylureas and metformin HCL have been proven in numerous clinical studies as combination is more effective than monotherapy using each drug in blood glucose control.

Also, new approaches are required in order to attain and maintain good glycaemic control over time and aggressive earlier introduction of combination therapy is being increasingly recommended over conventional stepwise strategies.

ELIGIBILITY:
Inclusion Criteria:

* Ages 30 to 75 at the time of screening visit
* Subjects with type 2 DM diagnosed for at least 3 months before screening
* Subjects with type 2 DM treated with monotherapy of 500mg ≤ metformin ≤ 1000mg for at lest 4 weeks prior to screening
* HbA1c ≥ 7.0% but ≤ 10.0% at the time of screening visit
* 21 kg/m2 ≤ BMI ≤ 40 kg/m2
* A negative pregnancy test for all females of childbearing potential
* Provision of signed and dated informed consent prior to any study procedures
* Ability and willingness to perform SMBG and record the data on the subject's diary

Exclusion Criteria:

* A history of acute metabolic complications such as diabetic ketoacidosis or hyperosmolar nonketotic coma within 3 months before screening
* Current therapy with anti-hyperglycemic agents (except metformin) use in the 4 weeks (8 weeks in case of thiazolidinedione) before screening
* Concomitant treatment prohibited during the study period

  * Any oral hypoglycemic agent other than glimepiride, metformin HCl, and fixed-dose combination of glimepiride and metformin HCl
  * Any insulin therapy over 7 days consecutively or intermittently in order to treat acute metabolic decompensation or systemic infection during the study
  * Intermittent use of systemic corticosteroids or large dose of inhaled steroids
* Subjects with clinically significant renal (serum creatinine level > 1.5 mg/dL in male and > 1.4 mg/dL in female) or hepatic disease (ALT and AST > 2x ULN)
* Clinically significant laboratory abnormality on screening labs or any medical condition that would affect the completion or outcome of the study in the opinion of the investigator and/or sponsor;
* Pregnant or lactating females
* History of drug or alcohol abuse
* Subjects who have a history of noncompliance with regards to follow-up medical care
* Subjects with known hypersensitivity to glimepiride, metformin HCL
* Night-shift workers
* Treatment with any investigational product in the last 3 months before study entry
* Others; subjects who have participated in this study

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2007-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Adjusted mean changes in HbA1c from baseline to the last visit | 12~24 weeks

SECONDARY OUTCOMES:
Adjusted mean changes in FPG from baseline to the last visit | 12~24 weeks
Response rate based on HbA1c and FPG levels measured at the last visit | 12~24 weeks
Frequency with hypoglycemic episode | 12~24 weeks
Adverse event | 12~24 weeks
Abnormal change from baseline in clinical laboratory | 12~24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dong Seob CHOI, Principal Investigator — Korea University Anam Hospital
Locations (1):
- Handok Pharmaceuticals, Co., LTD, Seoul, South Korea

REFERENCES:
- [Derived] Kim HS, Kim DM, Cha BS, Park TS, Kim KA, Kim DL, Chung CH, Park JH, Jang HC, Choi DS. Efficacy of glimepiride/metformin fixed-dose combination vs metformin uptitration in type 2 diabetic patients inadequately controlled on low-dose metformin monotherapy: A randomized, open label, parallel group, multicenter study in Korea. J Diabetes Investig. 2014 Nov;5(6):701-8. doi: 10.1111/jdi.12201. Epub 2014 Mar 16. PMID 25422771